CLINICAL TRIAL: NCT01784367
Title: Extracorporeal Lung Assist to Avoid Intubation in Patients Failing Noninvasive Ventilation for Acute Hypercapnic Respiratory Failure
Brief Title: Extracorporeal Lung Assist to Avoid Intubation in Patients Failing Noninvasive Ventilation for Hypercapnic ARF
Acronym: ECLAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Stefan Kluge, PD Dr. Stefan Kluge, Universitätsklinikum Hamburg-Eppendorf
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PV4190
Record Dates: First submitted 2013-01-30; First posted 2013-02-05 (Estimated); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-02

CONDITIONS: Hypercapnia; Respiratory Insufficiency
Keywords: Hypercapnia; noninvasive ventilation; acute respiratory failure; endotracheal intubation; invasive mechanical ventilation
MeSH Terms: conditions — Hypercapnia; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECLA-group (Experimental): Treatment with a pump driven, venovenous extracorporeal lung assist
  Interventions: Device: vv-ECCO2R (Novalung GmbH, Germany)

INTERVENTIONS:
Device: vv-ECCO2R (Novalung GmbH, Germany) — Treatment with the extracorporeal lung assist (ECLA) The ECLA is a pump driven (centrifugal pump) venovenous circuit, which removes carbon dioxide from the patients blood by means of a membrane through which the patients blood runs on the one side of the membrane and sweep gas on the other side removing the patient´s carbon dioxide. Blood flow range from 0.5 to 4.5 l/min and sweep gas flow between 1 and 10 l/min. At blood flows of 2 l/min and higher the device also oxygenates the patients blood. The diameter and length of cannulas and the sites of venous insertions are left to the decision of the treating physician. Cannulas are inserted in seldinger technique under sterile conditions. Function and patency of the extracorporeal circuit requires mild therapeutic anticoagulation.

SUMMARY:
The study´s intention is to evaluate the feasibility, safety and effectiveness of a pump driven extracorporeal device for removal of carbon dioxide from the blood in oder to avoid intubation and invasive mechanical ventilation in patients with acute respiratory failure retaining carbon dioxide due to the failure of their ventilatory muscle pump and not responding to prior non-invasive mask ventilation.

DETAILED DESCRIPTION:
The study´s intention is to evaluate the feasibility, safety and effectiveness of a pump driven extracorporeal device for removal of carbon dioxide from the blood in oder to avoid intubation and invasive mechanical ventilation in patients with acute respiratory failure retaining carbon dioxide due to the failure of their ventilatory muscle pump and not responding to prior non-invasive mask ventilation. Since intubation with subsequent (prolonged) invasive mechanical ventilation is associated with considerable side effects this new strategy has the potential to improve overall clinical outcome in this selected patient group.

ELIGIBILITY:
Inclusion Criteria:

* acute or acute-on-chronic hypercapnic respiratory insufficiency (pH ≤ 7,35, PaCO2 > 45 mmHg)
* failure of noninvasive ventilation
* fulfilling criteria for endotracheal intubation

Exclusion Criteria:

* under 18 years of age
* prior inclusion in other interventional study
* pregnancy
* heparin allergy or heparin-induced thrombocytopenia type 2
* on home non-invasive ventilator
* "Do not resuscitate" order or moribund condition
* life expectancy less than 6 months
* no informed consent available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kluge, MD, Principal Investigator — Department of Intensive Care Medicine, University Medical-Center Hamburg-Eppendorf
Locations (1):
- Department of Intensive Care Medicine, University Medical-Center Hamburg-Eppendorf (plus 10 further centres in Germany, Austria and the Netherlands), Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kluge S, Braune SA, Engel M, Nierhaus A, Frings D, Ebelt H, Uhrig A, Metschke M, Wegscheider K, Suttorp N, Rousseau S. Avoiding invasive mechanical ventilation by extracorporeal carbon dioxide removal in patients failing noninvasive ventilation. Intensive Care Med. 2012 Oct;38(10):1632-9. doi: 10.1007/s00134-012-2649-2. Epub 2012 Jul 27. PMID 22836139
- [Result] Braune S, Sieweke A, Brettner F, Staudinger T, Joannidis M, Verbrugge S, Frings D, Nierhaus A, Wegscheider K, Kluge S. The feasibility and safety of extracorporeal carbon dioxide removal to avoid intubation in patients with COPD unresponsive to noninvasive ventilation for acute hypercapnic respiratory failure (ECLAIR study): multicentre case-control study. Intensive Care Med. 2016 Sep;42(9):1437-44. doi: 10.1007/s00134-016-4452-y. Epub 2016 Jul 25. PMID 27456703
- See also: Department of principal investigator — http://www.uke.de

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: The historical controls were patients with acute hypercapnic respiratory failure refractory to NIV who were treated with IMV. The matching criteria were main diagnosis, age, SAPS-II score and pH.
Period: Overall Study
Arm/Group | ECLA-group | Control Group
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ECLA Group: Treatment with a pump driven, venovenous extracorporeal lung assist
  vv-ECCO2R (Novalung GmbH, Germany): Treatment with the extracorporeal lung assist (ECLA) The ECLA is a pump driven (centrifugal pump) venovenous circuit, which removes carbon dioxide from the patients blood by means of a membrane through which the patients blood runs on the one side of the membrane and sweep gas on the other side removing the patient´s carbon dioxide. Blood flow range from 0.5 to 4.5 l/min and sweep gas flow between 1 and 10 l/min. At blood flows of 2 l/min and higher the device also oxygenates the patients blood. The diameter and length of cannulas and the sites of venous insertions are left to the decision of the treating physician. Cannulas are inserted in seldinger technique under sterile conditions. Function and patency of the extracorporeal circuit requires mild therapeutic anticoagulation.
- Control Group: Control patients were identified and their data retrospectively collected from a large patient database at the principal study centre. The control patients had also been admitted to Intensive Care Unit with hypercapnic ventilatory failure and subsequently failed non-invasive ventilation (NIV) treatment followed by intubation and invasive mechanical ventilation. Matching criteria for the historical controls were acute diagnosis leading to hypercapnic respiratory failure, age (±10), SAPS-II score (±6) on ICU admission and pH (±0.06) at the time of NIV failure.
- Total: Total of all reporting groups
Arm/Group | ECLA Group | Control Group | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 15 | 15 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67 [51 to 83] | 68 [55 to 82] | 67 [51 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 12 | 13 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 25 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 21 | 25 | 46
  Netherlands | 2 | 0 | 2
  Austria | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Need for Intubation for Invasive Mechanical Ventilation
Description: The number of patients in the ECLA-group who had to be intubated and mechanically ventilated under the given criteria for inclusion and exclusion is collected. Since every patient in the matched control group was intubated, the comparison of the groups shows whether the use of a pump-driven venovenous extracorporeal lung assist can reduce the frequency of intubation and mechanical ventilation.
Time Frame: 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | ECLA-group | Control Group
Number analyzed (Participants) | 25 | 25
Participants | 11 | 25

2. Secondary Outcome: Length of Non-invasive Ventilation
Description: The duration of non-invasive ventilation up to day 90 is used to evaluate the respiratory outcomes of ECLA versus invasive mechanical ventilation.
Time Frame: 90 days
Population: As the control group receives 100% invasive mechanical ventilation by definition, this group is not analysed.
Measure: Mean (Full Range); unit: days
Arm/Group | ECLA-group | Control Group
Number analyzed (Participants) | 25 | 0
days | 4.6 [0 to 90] |

3. Secondary Outcome: Complication Rates
Description: Major complication associated with the pump driven extracorporeal lung assist device or with non-invasive or invasive mechanical ventilation or any associated treatments during the observational period
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | ECLA-group | Control Group
Number analyzed (Participants) | 25 | 25
Participants | 11 | 2

4. Secondary Outcome: Length of Invasive Mechanical Ventilation if Intubated
Description: Describes the length of invasive mechanical ventilation in days, in case intubation and mechanical ventilation became necessary
Time Frame: 90 days
Measure: Mean (Full Range); unit: days
Groups:
- Control Group: Matched historical control group
Arm/Group | ECLA-group | Control Group
Number analyzed (Participants) | 25 | 25
days | 8.3 [0 to 90] | 13.7 [1.0 to 90]

5. Secondary Outcome: Length of Stay in ICU
Description: Describes the length of stay in ICU
Time Frame: 90 days
Measure: Mean (Full Range); unit: days
Arm/Group | ECLA-group | Control Group
Number analyzed (Participants) | 25 | 25
days | 28.9 [0 to 90] | 24.0 [0 to 90]

6. Secondary Outcome: Mortality
Description: Comparison of 90-day mortality between the study arms. Seven patients died in each of the two arms after 90 days, so the stated values are correct.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | ECLA-group | Control Group
Number analyzed (Participants) | 25 | 25
Participants | 7 | 7

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | ECLA-group | Control Group
All-Cause Mortality (participants affected / at risk) | 7/25 | 7/25
Serious Adverse Events (participants affected / at risk) | 11/25 | 2/25
Other Adverse Events (participants affected / at risk) | 4/25 | 8/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECLA-group (N=25) | Control Group (N=25)
bleeding (Blood and lymphatic system disorders) | 11 (14) | 2 (2) — major bleeding
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECLA-group (N=25) | Control Group (N=25)
minor bleeding (Blood and lymphatic system disorders) | 4 (10) | 8 (10)

LIMITATIONS AND CAVEATS:
An important methodological limitation of our study is that the criteria used to define "NIV failure" and "indication for intubation" in the ECCO 2R group left a degree of subjective clinical judgement to the attending intensivist.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes